CLINICAL TRIAL: NCT01643720
Title: Emotion Regulation in Preschoolers With Autism and Their Parents
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC1013010kCTIL
Record Dates: First submitted 2012-07-04; First posted 2012-07-18 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2013-09

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva used for cortisol and oxytocin extraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorders: Children with Autism Disorders and their parents
- Typically Developing: Typically Developing children and their parents

SUMMARY:
In the proposed study, the investigators would like to investigate the emotion regulation (ER) strategies children with Autism Spectrum Disorders (ASD) demonstrate, and the influence parents have on their children's ER. More specifically, the investigators would like to examine what are the ER mechanisms that parents use, what mechanisms of self regulation children with autism internalize, and how parents support and improve the ER capabilities of their child with ASD. These will be studied in a behavioral level, using micro-analysis of parent-child interaction, and in a physiological level, using indexes of stress control and affiliation. In addition, in order for parental ER support to be effective, it is important to consider more innate neuro-developmental difficulties children with ASD demonstrate that strongly affect their ability to regulate themselves. These include sensory regulation difficulties, temperament, attention disorders and poor executive functioning.

Hypotheses:

1. ER strategies used by children with ASD will be more poorly developed and less effective, compared to those of children in the control groups.
2. Difficult temperament and sensory regulation difficulties will hamper ER in children with ASD.
3. ER strategies of parents of children with ASD will be more poorly developed and less effective than those of parents in the control groups.
4. Good parental self-ER and parental attunement to the child will be predictive of improved ER in children with ASD, and in parent-child synchrony, both in the behavioral and in the physiological levels.

ELIGIBILITY:
Inclusion Criteria:

* For the study group:Children diagnosed with ASD
* For the comparison group:Children with typical development

Exclusion Criteria:

* For the study group:Non verbal children.
* For the comparison group: Any major developmental disability.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants in the study group will be recrutied from psychiatric clinics, after a diagnosis of ASD has been made, and from special education kindergartens.
  participants in the comparison group will be recruited by adds suggesting participiation in the study that were published in variose cities and on the internet.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Emotion regulation(ER)strategies during emotion eliciting episodes | During a 2hr home visit, while the child interacts with the parent
  The Frequency,duration and percentage of ER behaviors presented by the child and the parent will be coded microanalytically using computerized coding system: The Observer, Noldus Co., Waggeniggen, The Netherlands

SECONDARY OUTCOMES:
Salivary hormone levels: Cortisol and Oxytocin of both parent and child | collected 4 times during the assessment meeting, from both child and parent.
  Changes in salivary Cortisol amd Oxytpcin levels over 3 time points during the home visit, before and after emotionally arousing activities. Collected from both parent and child.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Laor, MD, Study Chair — Brill Mental Health Center, Ramat Chen, Israel; Ofer Golan, PhD, Study Director — Department of Psychology, Bar-Ilan University, Ramat-Gan, Israel; Ruth Feldman, PhD, Study Director — Department of Psychology, Bar-Ilan University, Ramat-Gan, Israel; Nathaniel Laor, MD, Principal Investigator — Brill Mental Health Center, Ramat Chen, Israel
Locations (1):
- Brill Mental Health Center, Tel Aviv, Israel